CLINICAL TRIAL: NCT04810351
Title: Fever of Unknown Origin (FUO) in Elderly Patients
Acronym: FUO
Status: Recruiting | Type: Observational
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Nathalie compté, Clinic head of geriatric unit, Universitair Ziekenhuis Brussel
Other Study IDs: UZCompte2
Record Dates: First submitted 2021-03-11; First posted 2021-03-22 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Fever of Unknown Origin
Keywords: FUO; Fever of unknown origin
MeSH Terms: conditions — Fever of Unknown Origin | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Younger 1: young patients ( 18-69 years old) with oral or rectal fever > 37°8 or tympanic fever > 37°2 or CRP > 30 mg/dl during more than one week but less than three weeks of hospital with appropriate intelligent standard inpatient or outpatient workup to rule out usual causes of fever
  Interventions: Other: observational study
- Older 1: old patients ( > 70 years old) with oral or rectal fever > 37°8 or tympanic fever > 37°2 or CRP > 30 mg/dl during more than one week but less than three weeks out of hospital with appropriate intelligent standard inpatient or outpatient workup to rule out usual causes of fever
  Interventions: Other: observational study
- Young 2: young patients (18-69 years old) with oral or rectal fever > 37°8 or tympanic fever > 37°2 or CRP > 30 mg/dl during more than 3 weeks with appropriate intelligent standard inpatient or outpatient workup to rule out usual causes of fever.
  Interventions: Other: observational study
- Older 2: old patients ( > 70 years old) with oral or rectal fever fever > 37°8 or tympanic fever > 37°2 or CRP > 30 mg/dl during 3 weeks with appropriate intelligent standard inpatient or outpatient workup to rule out usual causes of fever13 .
  Interventions: Other: observational study

INTERVENTIONS:
Other: observational study — There is no intervention. It is an observational study

SUMMARY:
Objective: Fever of unknown (FUO) origin remains challenging in geriatric patients. Geriatric patients have a blunted immune response responsible for altered fever mechanisms and immune cells responses. Consequently, FUO could be inappropriately named and could be changed in Inflammation of unknown origin (IUO) in this specific population. Furthermore, the studies of FUO in this group are (out)dated and the diagnostic methods have evolved achieving a better sensitivity and specificity. The aim of our study is to assess the spectrum of diseases responsible of FUO or IUO in elderly patients compared to younger patients and to define the diagnostic approach using new diagnostic investigations. The second aim of our study is to assess the usefulness of inflammatory markers, demographic data and comorbidity to differentiate the cause of FUO/IUO.

Design: Patients with FUO or IUO will prospectively be recruited at the geriatric unit and the internal medicine unit of the UZ hospital during four years. The demographic, social and medical data will be screened. All diagnostic methods will be described.

DETAILED DESCRIPTION:
Until today, diagnose of fever of unknown origin remains challenging in elderly patients. The presentation of the disease is often atypical and this can delay diagnose and treatment. Geriatric patients have a blunted immune response responsible for altered fever mechanisms. For example, thirty-two percent of geriatric patients presented an infection at the emergency service having no pyrexia or increased white blood cell count in the presence of an infection.

Consequently, the definition of FUO in older patients is different from younger patients. FUO in older patients is defined as tympanic or axillar fever > 37.2.0C, a rectal fever more than 37.50C or a change of > 1.3 centigrade from basal temperature during more than 3 weeks. Furthermore, the name FUO is probably not appropriate in this population and should be replaced with inflammation of unknown origin. However, Unger et al also proposed inflammation of unknown origin in a younger population.

Knockaert et al have shown that the causes of FUO are different in older patients compared to young patients. The causes of FUO are more frequently found in older patients (> 65 years old) compared to younger patients (87-95% and 79% respectively). One explanation is the atypical presentation of classic diseases in geriatric patients. Infection, multi-system diseases and neoplasms were the most prevalent causes. These studies are old and the sensitivity and specificity of the diagnostic methods used presently, such as FDG-Pet-CT, have changed. The spectrum of diseases responsible of FUO or IUO in older patients could therefore have changed since the Knockaert studies. These new diagnostic methods allow better diagnose but also faster diagnose. Consequently the definition of FUO can become obsolete in the field of the duration of the fever.

Materials and Methods

The design of the study is an observational prospective study which will start in juli 2021 until open date in function of the number of included patient (at least 50 patients in both groups).

Patients will be recruited at the geriatric unit and internal medicine unit or geriatric outpatient clinic or internal medicine outpatient clinic of UZ Brussel and will be followed during one year.

The outpatient clinic patients will be recruited during the consultation; the patients who are hospitalized will be recruited during the first week of hospitalization.

The exclusion criteria are the impossibility to have an informed consent from the patient of a representative of the patient. Neutropenia, HIV or nosocomial fever of unknown origins are excluded. Immunodepressed patients are also excluded.

Patients:

All subjects will be screened for underlying illnesses by direct questioning, medical archives and blood sampling. Social evaluation will include determination of age, gender, home (private versus institution), and marital status. Clinical data will comprise: smoking and alcohol habits, old work, hobbies, travel, animal's owner, pneumococcal and influenza vaccine status, allergy, Body mass index (BMI), medical history, current treatment and reasons for hospitalization, recent antibiotic or corticoid treatment. For the older patients (> 70 years old) we will perform a CGA to identify comorbidity and common geriatric conditions. The polypathology and the severity of the medical problems will be scored using the "Charlson comorbidity Index"15 and "Cumulative Illness Rating Scale-Geriatric" (CIRS-G). It is an instrument to quantify disease burden. It comprises a comprehensive review of medical problems of 14 organ systems. It is based on a 0 to 4 rating of each organ system. The "Geriatric Depression Scale" will be used to assess the probability of depressed mood (GDS-15) in 15 questions. The assessment of "Activities of Daily Living" (ADL) will be made by using Katz's scale. It includes the following items: bathing, dressing, transfer, toilet, continence and eating. Each task is graded on a 3-level scale (1 to 3 for Katz's scale), where lower levels represent the absence of dependence and upper level the maximal dependence for the task. Cognitive functions will be assessed using the "Mini Mental State Examination" (MMSE). Possible scores range from 0 to 30 points, with lower scores indicating impaired cognitive function. Nutritional status was assessed using the "Mini Nutritional Assessment" (MNA). A score ≥ 24 identifies patients with a good nutritional status. Scores between 17 and 23.5 identify patients at risk of malnutrition. These latter patients have not yet started to lose weight and do not show low plasma albumin levels but have lower protein-caloric intakes than recommended. A score < 17 indicates protein-caloric malnutrition. Pain will be assess using a visual analogical scale from 0 to 10 points.

Methods

All diagnostic method means from the standard care of the patients during the hospital stay performed for the assessment of the fever or inflammatory syndrome will be collected:

* biological analyses, (such as CRP, renal function, lever function, electrolytes, sedimentation rates, uric acid, TSH, vitamin B12, folic acid, 25(OH) vitamin D, hemoglobin, hematocrit, proteins, albumin, white blood cells and formula, creatinine clearance (Cockcroft and de Gault formula), autoimmune assessment, viral or bacterial serology,…
* urine analyses
* Bacterial culture or PCR, viral PCR test in body fluids.
* Pleural puncture
* Lumbar puncture
* body sonography
* body X-rays and tomography
* Pet Ct
* Temporal artery biopsy
* Tissue biopsy
* Bronchoscopy
* Laparoscopy
* Bone marrow aspirate
* ….

Statistics:

Description statistics will be used such as means, medians, standard deviation and interquartile ranges.

Confidentiality All data will be collected by the investigators. The data will be collected in a way that patient names will not appear in the database (Redcap) and that individual patients will not be recognized by the examination of the collected data. Each patients will receive a code to preserve the anonymization. This code is a nummer that will be record on a listing of patients participating to the study in KWS. The listing in KWS is recorded in the worklisting CGER and is named FUO. Each investigator will be responsible of the anonymization of his/her recruiting. The database will only be accessible by the investigators and protected in Redcap by a password. The database (Excel) will be saved on UZBrussel server (CGER) in a folder named FUO.

ELIGIBILITY:
Inclusion criteria

* fever during more than one week out of hospital or more than 3 weeks with an intelligent appropriate workup
* an inflammatory syndrome during more than one week out of hospital or more than 3 weeks out of hospital
* The exclusion criteria :
* no inform consent
* Age < 18 years old
* Neutropenia, HIV or nosocomial fever of unknown origins are excluded. Immunodepressed patients are also excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited at the geriatric unit and internal medicine unit or geriatric outpatient clinic of UZ Brussel and will be followed during one year.
  Cfr inclusion and exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
the spectrum of diseases responsible of FUO or IUO | through study completion, an average of 1 year
  The proportion of infectious diseases, of neoplasm, of multi system disease of pulmonary embolism or deep vein thrombosis, of intoxication door medication will be measured in both groups
definition of FUO | through study completion, an average of 1 year
  we would like to compare fever of unknown origin since three weeks with fever of unknown origin since one week
Diagnostic approach of FUO | through study completion, an average of 1 year
  To describe the diagnostic approach and compare these diagnostic test in young and old population.

SECONDARY OUTCOMES:
Factors which influence FUO | At baseline
  Univariate and multivariate analyses will be used to measure the influence of age (years), gender, marital status, current treatment, comorbidities, recent use of antibiotics or corticoïd, Comprehensive geriatric assesment (MMSE, MNA, Katz, Lawton, CIRS-G, Charlson Index, GDS) on the cause of fever of unknown origin in both groups.

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Compte, MD, PhD, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (1):
- UZ brussel, Brussels, Jette, Belgium

IPD SHARING:
Plan to Share IPD: No
No plan

REFERENCES:
- [Background] Norman DC. Fever in the elderly. Clin Infect Dis. 2000 Jul;31(1):148-51. doi: 10.1086/313896. Epub 2000 Jul 25. PMID 10913413
- [Background] Norman DC, Yoshikawa TT. Fever in the elderly. Infect Dis Clin North Am. 1996 Mar;10(1):93-9. doi: 10.1016/s0891-5520(05)70288-9. PMID 8698997
- [Background] Tal S, Guller V, Gurevich A. Fever of unknown origin in older adults. Clin Geriatr Med. 2007 Aug;23(3):649-68, viii. doi: 10.1016/j.cger.2007.03.004. PMID 17631239
- [Background] Tal S, Guller V, Gurevich A, Levi S. Fever of unknown origin in the elderly. J Intern Med. 2002 Oct;252(4):295-304. doi: 10.1046/j.1365-2796.2002.01042.x. PMID 12366602
- [Background] Norman DC, Wong MB, Yoshikawa TT. Fever of unknown origin in older persons. Infect Dis Clin North Am. 2007 Dec;21(4):937-45, viii. doi: 10.1016/j.idc.2007.09.003. PMID 18061083
- [Background] Vanderschueren S, Del Biondo E, Ruttens D, Van Boxelaer I, Wauters E, Knockaert DD. Inflammation of unknown origin versus fever of unknown origin: two of a kind. Eur J Intern Med. 2009 Jul;20(4):415-8. doi: 10.1016/j.ejim.2009.01.002. Epub 2009 Feb 1. PMID 19524186
- [Background] Knockaert DC, Vanneste LJ, Bobbaers HJ. Fever of unknown origin in elderly patients. J Am Geriatr Soc. 1993 Nov;41(11):1187-92. doi: 10.1111/j.1532-5415.1993.tb07301.x. PMID 8227892
- [Background] Woolery WA, Franco FR. Fever of unknown origin: keys to determining the etiology in older patients. Geriatrics. 2004 Oct;59(10):41-5. PMID 15508555
- [Background] Gafter-Gvili A, Raibman S, Grossman A, Avni T, Paul M, Leibovici L, Tadmor B, Groshar D, Bernstine H. [18F]FDG-PET/CT for the diagnosis of patients with fever of unknown origin. QJM. 2015 Apr;108(4):289-98. doi: 10.1093/qjmed/hcu193. Epub 2014 Sep 9. PMID 25208896
- [Background] Schonau V, Vogel K, Englbrecht M, Wacker J, Schmidt D, Manger B, Kuwert T, Schett G. The value of 18F-FDG-PET/CT in identifying the cause of fever of unknown origin (FUO) and inflammation of unknown origin (IUO): data from a prospective study. Ann Rheum Dis. 2018 Jan;77(1):70-77. doi: 10.1136/annrheumdis-2017-211687. Epub 2017 Sep 19. PMID 28928271
- [Background] Mardi D, Fwity B, Lobmann R, Ambrosch A. Mean cell volume of neutrophils and monocytes compared with C-reactive protein, interleukin-6 and white blood cell count for prediction of sepsis and nonsystemic bacterial infections. Int J Lab Hematol. 2010 Aug 1;32(4):410-8. doi: 10.1111/j.1751-553X.2009.01202.x. Epub 2009 Nov 16. PMID 19919621
- [Background] Fusco FM, Pisapia R, Nardiello S, Cicala SD, Gaeta GB, Brancaccio G. Fever of unknown origin (FUO): which are the factors influencing the final diagnosis? A 2005-2015 systematic review. BMC Infect Dis. 2019 Jul 22;19(1):653. doi: 10.1186/s12879-019-4285-8. PMID 31331269